CLINICAL TRIAL: NCT03824678
Title: A Phase 1, Multicenter, Open-label Study to Evaluate the Pharmacokinetics of CC-220 in Subjects With Mild, Moderate, or Severe Hepatic Impairment Compared With Healthy Subjects
Brief Title: Evaluate the Pharmacokinetics of CC-220 in Subjects With Mild, Moderate, or Severe Hepatic Impairment Compared With Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-220-CP-007; U1111-1224-6064 (Registry Identifier: WHO)
Record Dates: First submitted 2019-01-09; First posted 2019-01-31 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Hepatic Impairment; Healthy Volunteers
Keywords: Hepatic impairment; Healthy Subjects; CC-220; Pharmacokinetics
MeSH Terms: interventions — iberdomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of CC-220 (Experimental): All subjects will receive one 1-mg CC-220 capsule administered orally with approximately 240 mL of non-carbonated, room temperature water, and administered by trained clinical staff.
  Interventions: Drug: CC-220

INTERVENTIONS:
Drug: CC-220 — CC-220

SUMMARY:
This is a multicenter, open-label study to assess the PK of a single 1-mg oral dose of CC-220 in subjects with mild, moderate, and severe hepatic impairment, and in matched healthy control subjects with normal hepatic function.

Degree of hepatic impairment will be determined during the Screening period by the subject's score according to Child-Pugh Classification Criteria

DETAILED DESCRIPTION:
Subjects will be enrolled in Groups 1 through 5 as follows:

* Group 1: Approximately 8 male or female subjects with mild hepatic impairment (with a Child Pugh score of ≥ 5 to ≤ 6) will be enrolled in Group 1.
* Group 2: Approximately 8 male or female subjects with moderate hepatic impairment (with a Child Pugh score of ≥ 7 to ≤ 9) will be enrolled in Group 2.
* Group 3: Approximately 8 male or female subjects with severe hepatic impairment (with a Child Pugh score of ≥ 10 to ≤ 13) will be enrolled in Group 3.
* Group 4: Approximately 8 healthy male or female subjects with normal hepatic function will be enrolled in Group 4. Subjects in Group 4 will be matched to subjects in Group 2 with respect to sex, age (± 10 years), and weight (± 13.6 kg [30 pounds]).
* Group 5: Approximately 8 healthy male or female subjects with normal hepatic function will be enrolled in Group 5. Subjects in Group 5 will be matched to subjects in Group 3 with respect to sex, age (± 10 years), and weight (± 13.6 kg [30 pounds]).

Subjects with mild, moderate, and severe hepatic impairment and subjects with normal hepatic function may start the study in parallel.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy all of the following criteria to be enrolled in the study:

1. Subject must understand and voluntarily sign an Informed Consent Form (ICF) prior to any study-related assessments/procedures being conducted.
2. Subject is willing and able to adhere to the study visit schedule and other protocol requirements, including the restrictions.
3. Subject is a male or female ≥ 18 and ≤ 70 years of age at the time of signing the ICF.
4. Subject has body mass index (BMI) ≥ 18 and ≤ 40 kg/m2 at Screening.
5. Subject agrees to abide by the requirements and restrictions outlined in the CC-220 Pregnancy Prevention Plan for Subjects in Clinical Trials.
6. Female subjects NOT of childbearing potential must:

   a. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before Screening, or postmenopausal (defined as 24 consecutive months without menses before Screening, with a follicle-stimulating hormone [FSH] level of > 40 IU/L at Screening).
7. Females of childbearing potential (FCBP)1 must have a negative pregnancy test at the Screening and baseline visits. All FCBP must use two effective birth control methods at the same time (for example: birth control pills, condoms, etc.) or practice complete abstinence from sexual contact with a man beginning 28 days before starting study treatment, throughout the entire duration of study treatment and at least 28 days after the end of study treatment with CC-220. The 2 methods of reliable contraception must include 1 highly effective method and 1 additional effective (barrier) method; options are described below:

   Examples of highly effective methods: intrauterine device; hormonal (birth control pills, injections, implants, levonorgestrel-releasing intrauterine system, medroxyprogesterone acetate depot injections, ovulation inhibitory progesterone-only pills [eg, desogestrel]); tubal ligation; or partner's vasectomy.

   AND Examples of additional effective methods: Male condom, diaphragm, or cervical cap.
8. Male subjects must:

   a. Practice true abstinence2 (which must be reviewed on a monthly basis, as applicable, and source documented) or agree to use a barrier method of birth control (condoms not made out of natural [animal] membrane [latex condoms are recommended]) during sexual contact with a pregnant female or FCBP while participating in the study, and for at least 90 days after the dose of IP, even if he has undergone a successful vasectomy.
9. Subject has clinical laboratory safety test results that are within normal limits or acceptable to the Investigator.
10. Subject is afebrile (febrile is defined as ≥ 38°C or 100.4°F), with sitting systolic blood pressure ≥ 90 and ≤ 160 mm Hg, sitting diastolic blood pressure ≥ 50 and ≤ 100 mm Hg, and pulse rate ≥ 40 and ≤ 100 beats per minute at Screening.

    Each subject with mild, moderate, or severe hepatic impairment must also meet all of the criteria listed below for entry:
11. Subject has mild, moderate, or severe hepatic impairment or cirrhosis due to chronic hepatic disease and/or prior alcohol abuse.
12. Subject has creatinine less than or equal to 1.5 x ULN.
13. Subject has mild (Group 1), moderate (Group 2), or severe (Group 3) hepatic impairment as defined by Child-Pugh score.

    * Group 1 subjects (mild hepatic impairment) are required to have documentary confirmation of the diagnosis of liver impairment made by biopsy, laparoscopy, or ultrasound with a Child-Pugh score of ≥ 5 to ≤ 6 at Screening.
    * Group 2 subjects (moderate hepatic impairment) are required to have documentary confirmation of the diagnosis of liver impairment made by biopsy, laparoscopy, or ultrasound with a Child-Pugh score of ≥ 7 to ≤ 9 at Screening.
    * Group 3 subjects (severe hepatic impairment): if biopsy, laparoscopy, or ultrasound is not performed prior to Screening, subjects can be included only if they have chronic liver disease and objective evidence of portal hypertension (ascites diagnosed by imaging or varices), with a Child-Pugh score ≥ 10 and ≤ 13 at Screening.

    Subjects should be enrolled into the group corresponding to the Child-Pugh classification score that most accurately reflects the most severe hepatic disease classification within the past 6 months (based on past medical history or PE observation).

    Note: If a Child-Pugh score was previously calculated and documented in the last 6 months, and it is more severe than the one calculated at Screening, then that previous value may be used for study entry purposes. If the Screening Child-Pugh score is more severe, then it will be used. If no score was calculated in the 6 months prior to Screening, then the score obtained at Screening will be used. Adequate documentation should be provided to substantiate the Child-Pugh score assigned to each subject.
14. Subject must be medically stable for at least 1 month before Screening with clinically acceptable medical history, PEs, clinical laboratory results, vital signs, and 12-lead ECGs consistent with the underlying hepatic impairment condition, as judged by the Investigator.
15. Subject is stable on a concomitant medication regimen (defined as not starting a new medication[s] or a change in the dosage or frequency of the concomitant medication[s] within 7 days or 5 half-lives [whichever is longer] before dosing with CC-220).
16. Subject may be treated with diuretics for ascites; however, subjects with severe ascites at time of enrollment may only be included at the discretion of the Investigator with agreement of Celgene.
17. Subject may have a history of encephalopathy; however, they must be on stable treatment for at least 1 month prior to Screening and must not have had an acute severe encephalopathic episode in the 1 month prior to Screening.
18. Subject has a normal or clinically acceptable 12-lead ECG at Screening (QT interval corrected for heart rate using Fridericia's formula [QTcF] ≤ 480 msec).

    Each matched healthy subject must also meet all the criteria listed below for entry:
19. Subject is free of any CS disease that would interfere with the study evaluations and has not had any unstable CS illness within 3 months prior to Screening.
20. Subject has liver-related laboratory test results within the respective reference ranges or with clinically insignificant excursions therefrom as agreed by the Investigator and Celgene's Medical Monitor.
21. Subject must match a subject in Group 2 or 3, as needed, primarily with respect to sex, age (± 10 years) and weight (± 13.6 kg [30 pounds]). Group 4 subjects will be matched with subjects from Group 2, and Group 5 subjects will be matched with Group 3 subjects.
22. Subject is in good health as determined by past medical history, PEs, vital signs, ECG, and clinical laboratory results. Clinical laboratory results (ie, hematology, chemistry, and urinalysis) and 12-lead ECGs must be within normal limits or clinically acceptable as judged by the Investigator. In addition:

    1. If male, subject has a QTcF value ≤ 440 msec at Screening.
    2. If female, subject has a QTcF value ≤ 460 msec at Screening.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant and relevant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject at an unacceptable risk if the subject was to participate in the study.
3. Subject has any condition that confounds the ability to interpret data from the study.
4. Subject is pregnant or breastfeeding or plans to become pregnant during the study or within 28 days of dosing.
5. Subject was exposed to an investigational drug (new chemical entity) within 30 days preceding the dose administration, or 5 half-lives of that investigational drug, if known (whichever was longer).
6. Subject has consumed any medication known to be a moderate or strong CYP3A inducer (including St. John's wort) within 30 days prior to dosing. The Indiana University P450 Drug Interactions Flockhart Table™ may be consulted for a list of such medications.
7. Subject has consumed any medication known to be a moderate or strong CYP3A inhibitor within 7 days prior to dosing. The Indiana University P450 Drug Interactions Flockhart Table™ may be consulted for a list of such medications.
8. Subject has consumed grapefruit, grapefruit juice, or any other grapefruit-containing product or oranges, orange juice, or any other product containing and/or made from oranges within 7 days prior to dosing.
9. Subject has any surgical or medical condition(s) possibly affecting drug absorption, distribution, metabolism, and excretion, eg, bariatric procedure. Subjects with appendectomy and cholecystectomy may be included.
10. Subject has donated blood or plasma within 2 weeks before the dose administration to a blood bank or blood donation center.
11. Subject has a history of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual) within 2 years before the dose administration, or positive drug Screening test reflecting consumption of illicit drugs, unless the positive drug screen is due to prescription drug use that is approved by the Investigator and Celgene's Medical Monitor.
12. Subject has a history of alcohol abuse (as defined by the current version of the Diagnostic and Statistical Manual) within 1 year before the dose administration, or a positive alcohol screen.
13. Subject has a positive result to the test for human immunodeficiency virus (HIV) antibodies at Screening.
14. Subject smokes more than 10 cigarettes per day, or the equivalent in other tobacco products (self-reported).
15. Subject is part of the clinical staff personnel or a family member of the study site staff.
16. Subject has received immunization with a live or live attenuated vaccine within 1 month prior to administration of the dose of CC-220 or is planning to receive immunization with a live or live attenuated vaccine 1 month after administration of the dose of CC-220.
17. Subject is, for any reason, deemed by the Investigator to be inappropriate for this study, including a subject who is unable to communicate or to cooperate with the Investigator or the clinical staff.

    The presence of any of the following will exclude a hepatically impaired subject from enrollment:
18. Subject has a hepatic impairment score of 14 or 15 at Screening as defined by Child-Pugh.
19. Subject has current hepatic encephalopathy with time or place disorientation, somnolence, stupor, coma, no personality/behavior, rigidity, or hyperactive reflexes - or has had such within 1 month of Screening.
20. Subject has a history of hepatorenal syndrome or hemolysis.

    Matched healthy subjects will be excluded from entry if any of the criteria listed below are met:
21. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
22. Subject has a positive test result for any active hepatitis, or history of Hepatitis B or Hepatitis C.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic- AUC0-t | Up to approximately 5 days
  Estimation of AUC calculated from time zero to the last measured time point
Pharmacokinetic- AUC0-∞ | Up to approximately 5 days
  Estimation of AUC calculated from time zero to infinity
Pharmacokinetic- Cmax | Up to approximately Day 1
  Estimation of observed maximum concentration
Pharmacokinetic- Tmax | Up to approximately Day 1
  Estimation of time to Cmax
Pharmacokinetic- t½ | Up to approximately 5 days
  Estimation of terminal elimination half-life
Pharmacokinetic- CL/F | Up to approximately 5 days
  Estimation of apparent clearance of drug from plasma after extravascular administration
Pharmacokinetic- Vz/F | Up to approximately 5 days
  Estimation of apparent volume of distribution during the terminal phase

SECONDARY OUTCOMES:
Adverse Event(s) | From consent to 28 days after the dose of IP
  Number of subjects with adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Alice Wang, MD, Study Director — Celgene
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Orlando Clinical Research Center OCRC, Orlando, Florida
  - The Texas Liver Institute, San Antonio, Texas